CLINICAL TRIAL: NCT04046952
Title: Radial Hemostasis is Facilitated With a Potassium Ferrate Hemostatic Patch (Statseal): the Randomized Controlled Statseal With TR Band Assessment Trial (STAT) II
Brief Title: Comparing TR Band to Statseal in Conjunction With TR Band II
Acronym: Statseal II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis at 50% of planned enrollment met prespecified critieria.
Sponsor: VA Long Beach Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arnold Seto, VA Long Beach Chief of Cardiology, Director of Interventional Cardiology Research, VA Long Beach Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRB 1843; NCT03116438 (obsolete NCT alias)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Arterial Occlusion; Cardiovascular Diseases; Atherosclerosis; Hematoma; Anticoagulant-induced Bleeding; Coronary Artery Disease
Keywords: Radial Artery Occlusion; Time to Hemostasis; Statseal; TR Band; cardiac catheterization; transradial catheterization; percutaneous coronary intervention
MeSH Terms: conditions — Arterial Occlusive Diseases; Cardiovascular Diseases; Atherosclerosis; Hematoma; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TR band only (Active Comparator): Patients will have a TR band applied over the arteriotomy site and inflated with 15-18ml of air. After aspirating and clearing the contents of the sheath, the radial sheath will be removed. The TR band will be deflated until bleeding occurs, and 2 ml of air will be reintroduced to provide hemostasis. Patent hemostasis will be documented with plethysmography and oximetry as described below within 5 minutes after band application and removal, and within 30 min of discharge or after 24 hours. The TR band will be left inflated and in place for 60 minutes following the procedure for all patients (regardless of diagnostic or PCI procedure), after which full deflation attempts will commence.
  Interventions: Device: TR band only
- Statseal with TR Band (Experimental): Patients will have a Statseal Advance RAD (SS) disc applied after withdrawing the radial sheath 2-4 cm. A Tegaderm dressing will be applied to secure the disc position. The TR band will be applied over the SS disc with the center of the balloon (the green dot) over the center of the SS disc. The TR band will be inflated with 8cc of air (which is typically occlusive pressure), and the sheath removed. No deflation will occur immediately. After 20 minutes of pressure, 3 cc of air will be removed from the TR band. After an additional 40 minutes (60 minutes after procedure), the TR band will be completely deflated.
  Interventions: Device: Statseal with TR Band

INTERVENTIONS:
Device: Statseal with TR Band — Patients will have a Statseal Advance RAD (SS) disc applied after withdrawing the radial sheath 2-4 cm. A Tegaderm dressing will be applied to secure the disc position. The TR band will be applied over the SS disc with the center of the balloon (the green dot) over the center of the SS disc. The TR band will be inflated with 8cc of air (which is typically occlusive pressure), and the sheath removed. No deflation will occur immediately. After 20 minutes of pressure, 3 cc of air will be removed from the TR band. After an additional 40 minutes (60 minutes after procedure), the TR band will be completely deflated.
  Arms: Statseal with TR Band
Device: TR band only — Patients will have a TR band applied over the arteriotomy site and inflated with 15-18ml of air. After aspirating and clearing the contents of the sheath, the radial sheath will be removed. The TR band will be deflated until bleeding occurs, and 2 ml of air will be reintroduced to provide hemostasis. Patent hemostasis will be documented with plethysmography and oximetry as described below within 5 minutes after band application and removal, and within 30 min of discharge or after 24 hours. The TR band will be left inflated and in place for 60 minutes following the procedure for all patients (regardless of diagnostic or PCI procedure), after which full deflation attempts will commence.
  Arms: TR band only

SUMMARY:
The purpose of this clinical study is to compare how well two different devices for achieving hemostasis perform in patients undergoing transradial procedures. Both devices are approved by the FDA for this use, and have already been used by clinicians on patients undergoing transradial procedures. It is believed that the use of both devices in combination compared to the hemostasis band (TR band) alone will shorten the time that it takes to 'seal' the artery, resulting in a shorter period of time that you would need to wear the hemostasis band.

DETAILED DESCRIPTION:
This study is a physician initiated, prospective, observational, two arm, randomized study to be performed at experienced 'Radial First' centers. Patients having undergone successful radial catheterization will be enrolled in the study. Enrollment with continue at each site with an initial goal of 800 patients enrolled, with each center contributing a minimum of 50 patients. Study will be have a single interim analysis after 400 patients are enrolled for efficacy and safety and continuation of the study. Clinicians will perform the catheterization in accordance with local standard practice, with no minimum amount of anticoagulation required.

Unlike the pilot trial of this device, the present study will have an identical time to first deflation of 60 minutes between the two groups, and have a larger sample size to detect any excess risk of hematoma or radial artery occlusion. The study may also help demonstrate a relatively low rate of radial artery occlusion with a rapid deflation protocol, even at lower doses of unfractionated heparin than currently recommended.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing diagnostic angiography or PCI via the radial artery
* Patients with a Barbeau test prior to the procedure showing pattern A,B,or C.

Exclusion Criteria: any one of the following...

* Use of a radial sheath larger than 6 Fr (a 7Fr-in-6 Glidesheath Slender ® is allowed).
* Use of a hemostasis method or device besides the TR Band.
* Patients undergoing catheterization from the femoral, brachial, ulnar, or distal radial (snuffbox) artery approach.
* Use of an anticoagulant other than unfractionated heparin or bivalirudin.
* Any use of glycoprotein inhibitors or cangrelor.
* Use of sheathless guides.
* Any anticipated need for continued anticoagulation post-catheterization, including extended bivalirudin infusion.
* Any active treatment with oral anticoagulants continued during course of procedure.
* Presence of arteriovenous dialysis fistula in the ipsilateral arm.
* Any physical deformity or trauma / injury of either wrist that would prevent proper placement or function of the hemostasis band.
* Raynaud's syndrome or known peripheral vascular disease of the forearm.
* Inability of the patient to personally consent for the study. (no surrogate consent)
* History or presence of Radial Artery Occlusion.
* Barbeau test showing Pattern D.
* Cardiogenic shock or any clinical instability as assessed by the physician performing the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Veteran Affairs Long Beach, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data would be made available to other researchers upon request by email and coauthor credit.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Starting May 1, 2021 and for 3 years thereafter.
Access Criteria: Email and coauthor credit

REFERENCES:
- [Derived] Safirstein JG, Tehrani DM, Schussler JM, Reid N, Mukerjee K, Weber L, Liu H, Skenderian S, Simeon M, Yang T, Seto AH. Radial Hemostasis Is Facilitated With a Potassium Ferrate Hemostatic Patch: The STAT2 Trial. JACC Cardiovasc Interv. 2022 Apr 25;15(8):810-819. doi: 10.1016/j.jcin.2021.12.030. PMID 35450681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2019 through December 2020, 443 patients were enrolled at 3 centers in the United States. Percutaneous coronary interventions (PCI) comprised 27% of procedures.
Groups:
- Statseal With TR Band: Patients will have a Statseal Advance RAD (SS) disc applied after withdrawing the radial sheath 2-4 cm. A Tegaderm dressing will be applied to secure the disc position. The TR band will be applied over the SS pad with the center of the balloon (the green dot) over the center of the SS pad. The TR band will be inflated with 8cc of air (which is typically occlusive pressure), and the sheath removed. No deflation will occur immediately. After 20 minutes of pressure, 3 cc of air will be removed from the TR band. After an additional 40 minutes (60 minutes after procedure), the TR band will be completely deflated.
Period: Overall Study
Arm/Group | TR Band Only | Statseal With TR Band
Started | 220 | 223
Completed | 220 | 223
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TR Band Only | Statseal With TR Band | Total
Number analyzed (Participants) | 220 | 223 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11) | 68 (10) | 67.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 42 | 109
  Male | 153 | 181 | 334
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 220 | 223 | 443
Weight [Mean (Standard Deviation); unit: lbs] | 199 (52) | 203 (46) | 200 (49)
Hypertension [Count of Participants; unit: Participants] | 167 | 176 | 343
Hypercholesterolemia [Count of Participants; unit: Participants] | 163 | 176 | 339
Diabetes Mellitus [Count of Participants; unit: Participants] | 69 | 86 | 155
Tobacco use [Count of Participants; unit: Participants] | 17 | 14 | 31
Barbeau's Class A [Count of Participants; unit: Participants] — Barbeau's classification of adequacy of dual-circulation of the hand after compression of radial and ulnar artery and releasing ulnar artery. Class A: No damping of pulse tracing immediately after compression, Class B:Damping of pulse tracing, Class C:Loss of pulse tracing followed by recovery of pulse tracing within 2 minutes. Class D:Loss of pulse tracing without recovery within 2 minutes. A was considered normal and D was considered at highest risk for radial occlusion.
  Participants | 79 | 76 | 155
Weak Pulse (<2+) [Count of Participants; unit: Participants] — Operator's subjective evaluation of pulse, graded as 0 (absent), 1+ (weak), and 2+ (normal)
  Participants | 76 | 92 | 168

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis Using the Hemostasis Management System (HMS)
Description: Time to deflation for removal of the TR Band (or TR Band and Statseal) for each group was measured in minutes.
Time Frame: Within 30 minutes of discharge or 24 hours post procedure (± 1 hour), whichever occurs first.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TR Band Only | Statseal With TR Band
Number analyzed (Participants) | 220 | 223
minutes | 113 (56) | 66 (14)

2. Secondary Outcome: Percent of Patients With Radial Artery Occlusion (RAO)
Description: Radial artery occlusion was monitored for all participants using Barbeau's test and pulse oximetry.
Time Frame: Within 30 minutes of discharge or 24 hours post procedure (± 1 hour), whichever occurs first.
Population: all patients examined
Measure: Count of Participants; unit: Participants
Arm/Group | TR Band Only | Statseal With TR Band
Number analyzed (Participants) | 220 | 223
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | TR Band Only | Statseal With TR Band
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/223
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/223
Other Adverse Events (participants affected / at risk) | 18/220 | 10/223
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TR Band Only (N=220) | Statseal With TR Band (N=223)
Any hematoma (Blood and lymphatic system disorders) | 15 (15) | 9 (9)
Bleeding requiring intervention (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — any intervention beyond TR band reinflation
Radial artery occlusion (Blood and lymphatic system disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to smaller number of subjects analyzed. Inability to blind operator and clinical evaluator to presence of patch. Ultrasound evaluation not performed routinely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT04046952/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04046952/ICF_001.pdf